CLINICAL TRIAL: NCT06089148
Title: Value of New Mammography Techniques in Comparison to Dynamic Contrast-Enhanced MRI of the Breast in the Detection and Diagnosis of Breast Lesions
Brief Title: New Mammographic Techniques Versus MRI in Assessment of Breast Lesions
Acronym: CEDM&DBTVSMR
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Marwa A Haggag, DR (lectureur), Cairo University
Other Study IDs: 141014
Record Dates: First submitted 2023-10-02; First posted 2023-10-18 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-10

CONDITIONS: Breast Diseases
MeSH Terms: conditions — Breast Diseases | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- contrast enhanced mammography, tomosynthesis and MRI: CEDM and tomosynthesis versus MRI
  Interventions: Diagnostic Test: contrast enhanced digital mammography, tomosyntheis and MRI

INTERVENTIONS:
Diagnostic Test: contrast enhanced digital mammography, tomosyntheis and MRI

SUMMARY:
Value of New Mammography Techniques in Comparison to Dynamic Contrast-Enhanced MRI of the Breast in the Detection and Diagnosis of Breast lesions

DETAILED DESCRIPTION:
Combined use of contrast-enhanced digital mammography (CEDM), and digital breast tomosynthesis (DBT), may be a reasonable alternative to MRI.

ELIGIBILITY:
Inclusion criteria

1. Breast Imaging Reporting and Data System (BI-RADS) 3, 4, and 5 breast lesions.
2. Clinical indication for MRI breast imaging.
3. No histologically proven cancer before enrollment. Exclusion criteria

1. Pregnancy or possible pregnancy. 2. History of allergy to an iodinated contrast agent. 3. Renal impairment. 4. Contraindication for MRI examination

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: FEMALE
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
sensitivity, specificity of'tomosynthesis and contrast enhanced mammography and MRI breast are measured in assessment of breast lesions and their pre-operative assessment of breast cancer | 1year
  diagnostic

IPD SHARING:
Plan to Share IPD: Yes
study protocol
Supporting Information: Study Protocol, SAP
Time Frame: 1year
Access Criteria: http://www.medicine.cu.edu.eg/index.php/en/
URL: http://www.medicine.cu.edu.eg/index.php/en/

REFERENCES:
- Available data/document: Study Protocol: Cairo unversity — https://medicine.cu.edu.eg/index.php/en/postgraduate/32-research/161-research-ethics-committee — upon requirement